CLINICAL TRIAL: NCT05190757
Title: Supraglottic Airway Needed To Achieve Ventilation (SANTA)
Brief Title: Supraglottic Airway Needed To Achieve Ventilation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Klaus D. Torp, Principal Investigator, Mayo Clinic
Other Study IDs: 21-008655
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Airway Complication of Anesthesia; Difficult or Failed Intubation
MeSH Terms: interventions — Ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laryngeal Mask Airway
  Interventions: Other: Airway and Ventilation
- Face Mask
  Interventions: Other: Airway and Ventilation

INTERVENTIONS:
Other: Airway and Ventilation — Insertion of Laryngeal Mask airway for ventilation or use of Face Mask

SUMMARY:
The purpose of this research is to compare if insertion of laryngeal mask airway (LMA) vs. use of face mask, will reduce the time needed to achieve adequate ventilation prior to insertion of the breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35.
* Patients willing to participate and provide an informed consent.
* Patients scheduled to undergo an elective surgical procedure including laparoscopic or robotic that requires GETA.

Exclusion Criteria:

* Patients who require administration of succinylcholine for induction/intubation
* Patients with history of uncontrolled GERD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Successful ventilation | Up to 15 minutes during the initial period of intubation.
  Compare time needed to achieve ventilation

SECONDARY OUTCOMES:
Subjective criteria of difficult ventilation and intubation | Up to 30 minutes during the initial period of intubation

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Torp, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials